CLINICAL TRIAL: NCT02804256
Title: Biomarkers of Inherited Cardiovascular Conditions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/933/C
Record Dates: First submitted 2016-05-31; First posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-05

CONDITIONS: Cardiomyopathy; Ischemic Heart Disease
MeSH Terms: conditions — Cardiomyopathies; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For antibody studies, the investigators will invite 10 patients with phenotypes of interest (e.g. myocardial fibrosis or previous myocardial infarction) whom have consented to the biorepository to provide an additional 20mls (2 tablespoons).
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Blood Sample Collection — 10 patients with ICCs to provide a second blood sample (20mls - 2 tablespoons) on top of the samples that will be collected for the biorepository.

SUMMARY:
The National Heart Centre Singapore has recently created a biorepository that is IRB approved for the use in genetic studies: "molecular and imaging studies of cardiovascular health and disease (CIRB Ref: 2013/605/C)". This repository enables IRB approved projects within the National Heart Centre Singapore to access the samples for use in biomarker or genetic studies with consent from patients for these studies. The IRB approved biorepository process also allows for patients, when they have consented to this, to be approached for inclusion in additional studies at National Heart Centre Singapore.

In this study, the investigators will examine the genetic variation in genes known to cause inherited cardiac conditions and also look for circulating biomarkers (ICC) in 600 patients with ICC and in 500 patients with ischemic heart disease (e.g.IHD) who will be used as controls. Healthy controls will also be used (800) as they become available in the biorepository. All samples have already been collected in the NHCS biorepository.

These patients would have been recruited and consented to the biorepository. This will enable all to better understand heart disease in Singaporean patients. In addition, the investigators will invite a subset of 10 patients with ICCs to provide a second blood sample (20mls - 2 tablespoons) on top of the samples that will be collected for the biorepository. The second blood sample will be used for antibody biomarkers that will be developed in the basic science laboratories. These antibodies will be used to develop new biomarkers of human heart disease to improve human health.

DETAILED DESCRIPTION:
In young adults and children inherited cardiac conditions (ICCs) that affect cardiac structure and electrical activity, account for most cases of sudden cardiac death. Of the ICCs, SCD due to Brugada Syndrome is particularly prevalent in SE Asia where it causes early loss of life in young men. While there have been major advances in the treatment of coronary artery disease (CAD), heart failure (HF) and acute MI, it remains very difficult to identify individuals at risk of SCD due to ICCs even when these diseases run in families and/or the mutation is known. This, in large part, relates to our limited understanding of the effects of gene mutations on clinical phenotypes due to variation in mutation penetrance and expressivity. In Singapore, and SE Asia in general, the issue of mutation interpretation is very difficult, if not impossible, as population-specific variant annotation is limited or completely absent for the common ICC genes. In addition, while DNA variants are important other protein biomarkers in the heart and in the vessels may be equally important, and these remain completely unaddressed in all populations.The investigatorswill address these issue in cases and controls using advanced sequencing and informatics approaches and by generating novel antibody libraries using patient samples.

Overall, the research performed in this study will find new ways of diagnosing patients at risk of sudden death both in the hospital environment and also in the general population. This will enable effective screening and stratification of patients at risk of sudden death due to inherited causes or following myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ICC.
* Patients with available cardiac/ cardiovascular imaging.
* Patients with phenotypes of interest (e.g. myocardial fibrosis, previous infarction).
* Age ≥ 21 years and ≤ 80 years.

Exclusion Criteria:

* Patients with HIV or hepatitis B or hepatitis C.
* Patients with active autoimmune disease.
* Patients who are unable or unwilling to provide consent.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will use DNA samples from 600 patients with known ICC diseases (e.g. Brugada syndrome, long QT syndrome, hypertrophic and dilated cardiomyopathy) and 500 ischemic controls who have been recruited or will be recruited to the NHCS biorepository.
  For antibody studies, the investigators will invite 10 patients with phenotypes of interest (e.g. myocardial fibrosis or previous myocardial infarction) whom have consented to the biorepository to provide an additional 20mls (2 tablespoons).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2014-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Biomarkers of inherited cardiovascular conditions from genetic variation in genes known to cause inherited cardiac conditions. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A Cook, PHD, Principal Investigator — National Heart Centre Singapore
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No